CLINICAL TRIAL: NCT05586061
Title: A Prospective, Multicenter, Phase II Clinical Study of First-line Treatment for HER2 (human Epidermal Growth Factor Receptor 2) Positive Advanced Gastric Cancer with Disitamab Vedotin in Combination with Tirelizumab and S-1
Brief Title: First-line Treatment with RC48 Plus Tislelizumab and S-1(RCTS) in Advanced Gastric Cancer
Acronym: RCTS
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Qilu Hospital of Shandong University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RCTS
Record Dates: First submitted 2022-10-16; First posted 2022-10-19 (Actual); Last update posted 2025-02-07 (Actual); Status verified 2025-02

CONDITIONS: HER2-positive Gastric Cancer
MeSH Terms: interventions — disitamab vedotin; tislelizumab; S 1 (combination)

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- RC48 Plus Tislelizumab and S-1(RCTS) (Experimental): Disitamab Vedotin: 2.5mg/kg, ivdrip, d1, (every 3 weeks) Q3W； Tislelizumab: 200mg, ivdrip, d1, (every 3 weeks) Q3W； S-1: 40-60mg(according to patients' body surface area), po, bid, d1-14 and discontinued for 7 days in each cycle; until progressive disease (PD) or intolerable toxicity
  Interventions: Drug: Disitamab vedotin; Drug: Tislelizumab; Drug: S1

INTERVENTIONS:
Drug: Disitamab vedotin — Disitamab Vedotin: 2.5mg/kg, d1, ivdrip, (every 3 weeks) Q3W
  Other Names: RC48
Drug: Tislelizumab — Tislelizumab: 200mg, d1, ivdrip, (every 3 weeks) Q3W
  Other Names: BGB-A317
Drug: S1 — S-1: 40-60mg (according to patients' body surface area), po, bid, d1-14, discontinued for 7 days.

SUMMARY:
This is a prospective, single arm, multicenter phase II study aimed at evaluating the efficacy and safety of Disitamab Vedotin in Combination With Tirelizumab and S-1 as first-line treatment for patients with advanced HER2-positive gastric or gastroesophageal junction adenocarcinoma.

ELIGIBILITY:
Inclusion Criteria:

1. Aged18-75 years, gender is not limited;
2. Pathologically confirmed locally advanced gastric or gastroesophageal junction adenocarcinoma that is inoperable or has distant metastasis;
3. HER2 was detected as 2+or 3+ by immunohistochemistry（IHC） ;
4. Has at least 1 measurable lesion as determined by RECIST 1.1;
5. There is no systematic treatment in the past, or the patient has received neoadjuvant/adjuvant chemotherapy, but the disease progresses or relapses more than 6 months after the end of treatment;
6. Eastern Cooperative Oncology Group (ECOG) performance status of 0-1;
7. Adequate organ function:

   1. Bone marrow function: i. Hemoglobin count (HGB)≥80g/L; ii. Neutrophil count (NE)≥1.5×109/L; iii. White blood cell count (WBC)≥3.5×109/L; iv. Platelet count (PLT)≥100×109/L；
   2. Liver function: i. Serum total bilirubin (TBIL)≤1.5×ULN; ii. Alanine aminotransferase (ALT), aspartate aminotransferase (AST) and alkaline phosphatase (ALP)≤3×ULN, patients with liver metastasis≤5×ULN;
   3. Kidney function: Blood creatinine (Cr) ≤1.5×ULN or Cockcroft Gault formula ≥ 60 mL/min;
   4. Cardiac function: New York Heart Association (NYHA) classification<Grade 3; Left ventricular ejection fraction≥50%;
8. The life expectancy is at least 3 months;
9. Female of childbearing age must have taken reliable contraceptive measures or conducted a pregnancy test (serum or urine) within 7 days before enrollment, and the result is negative, and are willing to use appropriate methods of contraception during the trial period and 8 weeks after the last administration of the test drug; For male, they must agree to use appropriate methods of contraception during the trial and 8 weeks after the last administration of the trial drug;
10. Willing to join the study and signed an informed consent form (ICF) with good compliance and cooperation in follow-up.

Exclusion Criteria:

1. Allergy to any trial drug and its excipients, or serious allergy history, or contraindication of the trial drug;
2. Cardiovascular and cerebrovascular events that are not well controlled, such as:

   1. NYHA grade 2 or above heart failure;
   2. Unstable angina pectoris;
   3. Myocardial infarction occurred within 1 year;
   4. Supraventricular or ventricular arrhythmia with clinical significance needs treatment or intervention;
   5. Cerebral hemorrhage and cerebral infarction (except for lacunar cerebral infarction without symptoms and without treatment);
   6. Serious cardiovascular and cerebrovascular events occurred within 12 months;
   7. Uncontrolled hypertension, i.e. systolic blood pressure>140 mmHg or diastolic blood pressure>90 mmHg after single drug treatment;
   8. Patients with history of arterial thrombosis or deep vein thrombosis within 6 months before recruitment, or with evidence of bleeding tendency or medical history within 2 months before recruitment, regardless of the severity;
   9. Stroke event or transient ischemic attack occurred within 12 months before recruitment;
3. Has received systematic treatment with Chinese patent medicine or immunomodulatory drugs (including thymosin, interferon, interleukin, except for local use for ascites control) before the first administration within 2 weeks.
4. Have a history of interstitial lung disease, non-infectious pneumonia, pulmonary fibrosis, acute lung disease, or systemic disease with poor control (including but not limited to diabetes, hypertension, etc.);
5. Have a history of active immune deficiency or autoimmune diseases, including HIV positive test, or have other acquired or congenital immune deficiency diseases, or have a history of organ transplantation or autoimmune diseases;
6. Severe chronic or active infection requires systemic antibacterial, antifungal or antiviral treatment, including tuberculosis infection.Have a history of active tuberculosis infection ≥ 1 year before recruitment should also be excluded, unless proved has been completed appropriate treatment;
7. Brain metastasis or leptomeningeal metastasis;
8. Clinically significant pleural effusion, pericardial effusion or ascites should be drained for many times within 2 weeks before the first administration of the trial drug;
9. Has a second clinically detectable primary malignant tumor at the time of recruitment, or there were other malignant tumors in the past 5 years (except for fully treated skin basal cell carcinoma or cervical carcinoma in situ);
10. Any major surgery was performed ≤ 28 days before the first trial drug administration;
11. History of allogeneic stem cell transplantation or organ transplantation;
12. Duodenal ulcer, ulcerative colitis, intestinal obstruction and other gastrointestinal diseases at present; or other conditions that may cause gastrointestinal bleeding or perforation judged by the researchers; or history of intestinal perforation or fistula, but has not recovered after surgical treatment;
13. Live vaccine was inoculated within 4 weeks (inclusive) before the first administration of the trial drug, not including seasonal influenza vaccines but intranasal vaccine.
14. Has other factors that may lead to the forced termination of this trial according to the judgment of the investigator, such as other serious diseases (including psychological and mental diseases) requiring combined treatment, serious laboratory examination abnormalities, and family or social factors, which may affect the safety of the subject, or the collection of data and samples;
15. Participating in other therapeutic clinical studies or using research instruments within 4 weeks before the first administration;
16. Others conditions do not meet the inclusion according to the judgment of the investigator.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2023-02-10 (Actual); Primary Completion 2024-12-29 (Actual); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
objective response rate (ORR) | 6 months after the last subject participating in
  The proportion of subjects with complete response (CR) and partial response (PR) in total subjects

SECONDARY OUTCOMES:
progression-free survival (PFS) | 12 months after the last subject participating in
  Progression-free survival (PFS per RECIST 1.1) is defined as the time from the starting date of study drug to the date of first documentation of disease progression or death, whichever occurs first
overall survival (OS) | 12 months after the last subject participating in
  OS is defined as the time from the starting date of study drug to the date of death due to any cause.
disease control rate (DCR) | 12 months after the last subject participating in
  The proportion of subjects with complete response (CR) and partial response (PR) and stable disease(SD)in total subjects
duration of response (DOR) | 12 months after the last subject participating in
  DOR (per RECIST 1.1) is defined as the time from the date for first documented response of complete response (CR) or partial response (PR) to the date of first documented of disease progression or death, whichever occurs first.

CONTACTS AND LOCATIONS:
Overall Officials: Lian Liu, Doctor, Principal Investigator — Qilu Hospital of Shandong University
Locations (7):
- China (7):
  - Central Hospital Affiliated to Shandong First Medical University, Jinan, Shandong
  - Qilu Hospital of Shandong University, Jinan, Shandong
  - Shandong Provincial Hospital Affiliated to Shandong First Medical Universiry, Jinan, Shandong
  - The First Affiliated Hospital of Shandong First Medical University (Shandong Provincial Qianfoshan Hospital), Jinan, Shandong
  - The Affiliated Hospital of Qingdao University, Qingdao, Shandong
  - Qingdao Municipal Hospital (Group), Qingdao, Shandong
  - Yantai Yuhuangding Hospital, Yantai, Shandong